CLINICAL TRIAL: NCT05685979
Title: Evaluation of Cardiac Functions in Robotic-assisted Prostatectomy Surgery Performed Under Deep Trendelenburg Position
Brief Title: Evaluation of Cardiac Functions in Deep Trendelenburg Position
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ATADEK; 2022-20/05
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hemodynamic Instability; Cardiovascular Complication
Keywords: Deep Trendelenburg position; Robotic-assisted laparoscopic prostatectomy; Pressure recording analytical method; Transesophageal echocardiography; Cardiac cycle efficiency; Longitudinal Strain; Hemodynamic monitorization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing robotic-assisted laparoscopic prostatectomy in deep Trendelenburg position.: Patients with ASA( American Society of Anesthesiologists) physical status 1-3 who underwent robotic-assisted laparoscopic prostatectomy in deep Trendelenburg position.
  Interventions: Procedure: Robotic-assisted laparoscopic prostatectomy in deep Trendelenburg position.

INTERVENTIONS:
Procedure: Robotic-assisted laparoscopic prostatectomy in deep Trendelenburg position. — After general anesthesia induction, the patients were placed in the deep Trendelenburg position (at least 25°-45° upside down).

SUMMARY:
Robotic-assisted laparoscopic prostatectomy (RALP) is a surgical method with good short-term results and accepted as the gold standard because of its minimal invasiveness. The pneumoperitoneum and deep Trendelenburg position (at least 25°-45° upside down) required for RALP surgeries can cause significant pathophysiological changes in both the pulmonary and cardiac systems, as well as complicate hemodynamic management.

In this study, investigators aimed to determine the changes in the cardiovascular system during deep Trendelenburg position with the hemodynamic parameters monitored by the pressure record analytical method (PRAM) and the Longitudinal Strain measured with simultaneous transesophageal echocardiography.

DETAILED DESCRIPTION:
RALP is the gold standard surgical technique in prostate surgery. Many Robotic-laparoscopic surgical techniques also require the intraoperative deep Trendelenburg position. However, the possible side effects of the deep Trendelenburg position on the cardiovascular system during surgery are unknown. Although the Trendelenburg position is a life-saving maneuver in hypovolemic patients, it also carries undesirable risks. Although the increase in venous return is expected to protect the cardiac output (CO) in the deep Trendelenburg position, the increase in intrathoracic pressure due to the intraperitoneal pressure may cause deterioration in venous return and a decrease in CO . In addition, the changing heart configuration in the deep Trendelenburg position may also cause an increase in the workload of the heart. Therefore, the need to evaluate hemodynamic management with advanced monitoring techniques, including fluid therapy in the perioperative period, has arisen in patients undergoing RALP.

The pressure Recording Analytical Method (PRAM), is one of the most up-to-date monitoring methods designed for continuous CO measurement derived from the arterial pressure wave analysis, with a high signal sampling rate (1000 Hz). Many studies have shown that PRAM is a reliable monitoring method in major surgery. Cardiac Cycle Efficiency (CCE), which the PRAM method adds to our daily practice, is an index that defines hemodynamic performance in terms of energy consumption and efficiency. It can be expressed as the ratio of systolic energy performance to the total energy expenditure of the cardiac cycle and indicates the ability of the cardiovascular system to maintain homeostasis at different energy levels. However, data on how cardiac functions change in the deep Trendelenburg position are still limited.

In this study, investigators aimed to demonstrate the reliability of the CCE value through its correlation with the Longitudinal Strain (LS) by observing the effect of the deep Trendelenburg position in RALP surgeries on cardiac functions using PRAM and Transesophageal Echocardiography (TEE).

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society Of Anesthesiology physical status 1-3
* Underwent Robotic-assisted laparoscopic prostatectomy
* Patients with intra-arterial blood pressure monitoring before anesthesia induction.

  .Exclusion Criteria:
* Under 18 years of age
* Arrhythmia (atrial fibrillation, frequent premature beat)
* History of myocardial infarction in the last 3 months
* Heart failure
* Severe pre-existing lung disease
* Severe valvular heart disease
* Chronic renal disease on dialysis,

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with ASA (American Society Of Anesthesiology) physical status 1-3 who underwent RALP with intra-arterial blood pressure monitoring before anesthesia induction
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Cardiac cycle efficiency (CCE) was measured for evaluating cardiac performance | The duration of the measurement was defined from one minute before induction to the end of the surgery
  CCE(unit) indicates the ability of the cardiovascular system to maintain homeostasis at different energy levels. CCE was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy)
Longitudinal strain (LS) was measured for evaluating cardiac performance | LS was measured at supine position and 10 minute after trendelenburg position
  LS (%) is a parameter that shows the percentage of dimensional change that occurs in the heart muscle. It is an indicator of the systolic functions of the left ventricle. LS was calculated by intraoperative transesophageal echocardiography.
Longitudinal strain rate (LSR) was measured for evaluating cardiac performance | LSR was measured at supine position and 10 minute after trendelenburg position
  LSR (%) is a parameter that shows the rate of dimensional change that occurs in the heart muscle. It is an indicator of the systolic functions of the left ventricle. LSR was calculated by intraoperative transesophageal echocardiography.

SECONDARY OUTCOMES:
Stroke volume variation (SVV) was measured for evaluation of volume status | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Stroke volume variation (SVV,%), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SVV is a parameter used to asses cardiac preload and fluid responsiveness.
Pulse pressure variation (PPV) was measured for evaluation of volume status | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Pulse pressure variation (PPV,%) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). PPV is a parameter used to asses cardiac preload and fluid responsiveness.
Cardiac power output (CPO) was measured for evaluation of cardiac power reserve | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Cardiac power output (CPO, Watt) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CPO is a parameter used to asses cardiac reserve
Cardiac index (CI) was measured for evaluating cardiac flow | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Cardiac index (CI, L/min/m2), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CI is a parameter used to asses cardiac stroke volume
Dp/Dt was measured to assess cardiac systolic function | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Dp/Dt(mmHg/msn), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). Dp/Dt is a parameter used to asses cardiac contractility.
Systolic arterial pressure (SAP) was measured for evaluating perfusion pressure | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Systolic arterial pressure (SAP- mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SAP is a parameter used to assess the pressure of the arterial system during cardiac systole
Diastolic arterial pressure (DAP) was measured for evaluating perfusion pressure | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Diastolic arterial pressure (DAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). DAP is a parameter used to assess the pressure of the arterial system during cardiac diastole
Mean arterial pressure (MAP) was measured for evaluating perfusion pressure | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Mean arterial pressure (MAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). MAP is a parameter used to assess organ perfusion
Heart rate (HR) was measured for evaluating heart ritm | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Heart rate( HR, bpm) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). HR is a parameter used to assess the cardiac rate.
Systemic vascular resistance index (SVRI) was measured for evaluating peripheric vascular resistance | The duration of the measurement was defined from one minute before induction to the end of the surgery
  Systemic vascular resistance index (SVRI, dyn*s/cm5*m2) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SVRI is a parameter used to assess the resistance to blood flow offered by all of the systemic vasculatures, excluding the pulmonary vasculature.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porpiglia F, Morra I, Lucci Chiarissi M, Manfredi M, Mele F, Grande S, Ragni F, Poggio M, Fiori C. Randomised controlled trial comparing laparoscopic and robot-assisted radical prostatectomy. Eur Urol. 2013 Apr;63(4):606-14. doi: 10.1016/j.eururo.2012.07.007. Epub 2012 Jul 20. PMID 22840353
- [Background] Falabella A, Moore-Jeffries E, Sullivan MJ, Nelson R, Lew M. Cardiac function during steep Trendelenburg position and CO2 pneumoperitoneum for robotic-assisted prostatectomy: a trans-oesophageal Doppler probe study. Int J Med Robot. 2007 Dec;3(4):312-5. doi: 10.1002/rcs.165. PMID 18200624
- [Background] Lestar M, Gunnarsson L, Lagerstrand L, Wiklund P, Odeberg-Wernerman S. Hemodynamic perturbations during robot-assisted laparoscopic radical prostatectomy in 45 degrees Trendelenburg position. Anesth Analg. 2011 Nov;113(5):1069-75. doi: 10.1213/ANE.0b013e3182075d1f. Epub 2011 Jan 13. PMID 21233502
- [Background] Pawlik MT, Prasser C, Zeman F, Harth M, Burger M, Denzinger S, Blecha S. Pronounced haemodynamic changes during and after robotic-assisted laparoscopic prostatectomy: a prospective observational study. BMJ Open. 2020 Oct 5;10(10):e038045. doi: 10.1136/bmjopen-2020-038045. PMID 33020097
- [Background] Ruppert M, Lakatos BK, Braun S, Tokodi M, Karime C, Olah A, Sayour AA, Hizoh I, Barta BA, Merkely B, Kovacs A, Radovits T. Longitudinal Strain Reflects Ventriculoarterial Coupling Rather Than Mere Contractility in Rat Models of Hemodynamic Overload-Induced Heart Failure. J Am Soc Echocardiogr. 2020 Oct;33(10):1264-1275.e4. doi: 10.1016/j.echo.2020.05.017. Epub 2020 Aug 7. PMID 32778499
- [Background] Faragli A, Tanacli R, Kolp C, Abawi D, Lapinskas T, Stehning C, Schnackenburg B, Lo Muzio FP, Fassina L, Pieske B, Nagel E, Post H, Kelle S, Alogna A. Cardiovascular magnetic resonance-derived left ventricular mechanics-strain, cardiac power and end-systolic elastance under various inotropic states in swine. J Cardiovasc Magn Reson. 2020 Nov 30;22(1):79. doi: 10.1186/s12968-020-00679-z. PMID 33256761